CLINICAL TRIAL: NCT06512545
Title: Second Haploidentical Transplantation with Modified Regimen for Graft Failure After the First Allogeneic Stem Cell Transplantation
Brief Title: Modified Second Haplo-transplantation for Graft Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Prof., Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHB181-001
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Graft Failure; Stem Cell Transplant Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention arm (Experimental): second haploidentical stem cell transplantation
  Interventions: Other: second allogeneic stem cell transplantation

INTERVENTIONS:
Other: second allogeneic stem cell transplantation — 1. Change another donor if possible
  2. Conditioning regimen: fludarabine (30mg/m2/day, days -6 to -2 )/cyclophosphamide (1g/m2/day, days -5 to -4)/rabbit antithymocyte globulin (1.5mg/kg/day, days -4 to -2)
  3. GVHD prophylaxis: cyclosporine A (concentration 150-250ng/ml), mycophenolate mofetil (0.5g bid -3d to neutrophil engraftment)+anti CD25 monoAb (20mg, +1d, +8d, +15d)

SUMMARY:
Graft failure is a fatal complication following allogeneic stem cell transplantation where a second transplantation is usually required for salvage. We previously reported encouraging results with a novel Flu/Cy regimen. However, there are still around 20% patients developed delayed platelet recovery. We designed a modified regimen to further improve the hematopoietic reconstitution after second transplantation. This prospective, single-arm study aims to investigate the safety and efficacy of this modified regimen.

ELIGIBILITY:
Inclusion Criteria:

* 1.Primary disease: hematological malignancies(AML, CML, MDS, lymphoma, etc.); 2.Graft failure after first allogeneic stem cell transplantation; 3.Time from the first transplantation to the second transplantation is less than 180 days; 4. Age≥14 years.

Exclusion Criteria:

* 1. Active infections; 2. Active GVHD; 3. Organ dysfunction: hepatic injury (Tbil≥2ULN), renal injury (Cr≥1.5ULN), heart injury (EF%<50% or symptomatic heart failure); 4. Eastern Cooperative Oncology Group (ECOG) score>2; 5. Expected life time<30 days; 5. Patients could not cooperate; 6. Other situations that are considered inappropriate for enrollment by the investigators,

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Engraftment of neutrophils | 28 days after second transplantation
  Engraftment of neutrophils was defined as the first of 3 consecutive days when the absolute neutrophil count achieved 500/uL.

SECONDARY OUTCOMES:
Engraftment of Platelet | 100 days after second transplantation
  Platelet engraftment was defined as the first of 7 consecutive days that platelet counts ≥20 × 10^9/L in the absence of platelet transfusion
TRM at 28 day | 28 days after second transplantation
  treatment-related mortality(TRM) was defined as death from any cause other than relapse.
TRM at 100 day | 100 days after second transplantation
  treatment-related mortality (TRM) was defined as death from any cause other than relapse
GVHD | Participants will be followed for an expected average of 1 year
  Both acute and chronic GVHD was diagnosed and graded according to international criteria.
OS | Participants will be followed for an expected average of 1 year
  Overall survival (OS)
LFS | Participants will be followed for an expected average of 1 year
  Leukemia-free survival (LFS) was defined as the survival period with continuous CR.
CIR | Participants will be followed for an expected average of 1 year
  The cumulative incidence of relapse (CIR)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, M.D., Principal Investigator — Institute of Hematology, Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No